CLINICAL TRIAL: NCT05075902
Title: Effect of Aerobic Training on Hemodynamic, Metabolic and Climacteric Symptoms in Postmenopausal Women With Multimorbidity
Brief Title: Effect of Aerobic Training on the Health Parameters of Postmenopausal Women With Multimorbidity
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Juliene Gonçalves Costa, Principal Investigator Juliene Gonçalves Costa Dechichi, Federal University of Uberlandia
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CAAE: 12453719.1.0000.5152
Record Dates: First submitted 2021-08-25; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Multimorbidity; Multiple Chronic Conditions; Hypertension; Dyslipidemias
Keywords: aerobic training; multimorbidity; menopause; blood pressure; arterial stiffness
MeSH Terms: conditions — Multiple Chronic Conditions; Hypertension; Dyslipidemias | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental controlled trial with a 12-week aerobic training intervention in postmenopausal women with and without cardiometabolic multimorbidity. Participants were allocated into groups according to the amount of cardiometabolic diseases, with the Morbidity group (MORB) being composed of women with one or no chronic cardiometabolic disease and the Multimorbidity group with two or more chronic cardiometabolic diseases.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The Care Providers followed the standard of care for all participants during the training sessions, with a standardized approach such as: measuring the blood pressure of all participants before starting the training session, intensity control during training was done by zone of individualized heart rate, regardless of the group, presented in a spreadsheet without information about the group to which the patient was assigned. The outcomes assessor were not aware of the formation of groups and access only to the participants' codes, were objective and with generation of saved files for later conference by the Investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimorbidity Group (MULTI) (Experimental): Multimorbidity group is composed of post menopausal women with two or more chronic diseases cardiometabolic (Hypertension, diabetes, dislipidemias, obesity).
  Interventions: Behavioral: Aerobic training
- Morbidity Group (MORB) (Experimental): Morbidity group is composed of postmenopausal women with one or no chronic cardiometabolic disease (Hypertension, diabetes, dislipidemias, obesity)
  Interventions: Behavioral: Aerobic training

INTERVENTIONS:
Behavioral: Aerobic training — The program consists of aerobic exercise performed three times a week on non-consecutive days for 12 weeks at an intensity of 65% to 75% of the reserve heart rate. During the first 4 weeks of training, the exercise duration was 40 minutes (5' warm up + 30 minutes in the intensity zone + 5' cool down). From the fifth week onwards, there was only an increase in volume to 50 minutes in duration (5'warm-up + 40 minutes in the intensity zone + 5'warm-up). The aerobic fitness assessment was performed on a maximal effort ergospirometric treadmill under the supervision of a qualified physician, using the Bruce protocol (adapted) to assess cardiopulmonary capacity (to assess possible cardiovascular capacity that prevents the proposed training) and for individualized training prescription.
  Other Names: Aerobic physical exercise

SUMMARY:
People affected by multiple chronic diseases have a greater chance of hospitalization, longer hospital stays, worse general health, worse physical and mental function and lower functional capacity, with an average risk of 50% of functional decline with each additional condition. The frequency of multimorbidity is higher in older, inactive women, who live in urban areas in low- and middle-income countries, the most affected by multimorbidity. The practice of physical exercise is an important component in the prevention of multiple chronic diseases, in which lower levels of physical activity were associated with an increased prevalence of multimorbidity in women aged 16 to 24 years. And regardless of the presence of multimorbidity, engaging in a healthier lifestyle, including regular physical activity, was associated with up to 7.6 more years of life for women, improving the individual's general health status even when multimorbid.

The hypothesis is that multimorbid women have a worse general health status when compared to women without multimorbidity, but aerobic exercise will be able to improve health parameters in 12 weeks of training.

This is a quasi-experimental clinical trial with a 12-week aerobic training intervention in postmenopausal women with and without cardiometabolic multimorbidity. Participants were allocated into groups according to the amount of cardiometabolic diseases, with the Morbidity group (MORB) being composed of women with one or no chronic cardiometabolic disease and the Multimorbidity group (MULTI) with two or more chronic cardiometabolic diseases.

The assessments of arterial stiffness, 24-hour ambulatory pressure, blood pressure variability, heart rate variability, lipid and glucose profile, body composition and climacteric symptoms were performed before and after the training period.

The study was carried out at the Laboratory of Cardiorespiratory and Metabolic Physiology at the Faculty of Physical Education of the Federal University of Uberlândia, Uberlândia, Brazil and approved by the Ethics Committee for studies in humans (CAEE: 12453719.1.0000.5152). All participants signed a consent form. The experiments followed the principles of the Declaration of Helsinki.

The program consists of aerobic physical exercises performed three times a week on non-consecutive days for 12 weeks with an intensity of 65% to 75% of the reserve heart rate.

DETAILED DESCRIPTION:
The sample size was classified using the G * Power 3.1 software (University of Dusseldorf, Dusseldorf, Germany), adopting an α error of 5%, 80% power analysis, 0.5 correlation between repeated measures and a correction of non-sphericity of 1, in an F-family of intra-between analysis. Changes in serum triglycerides were evaluated as the primary study endpoint. The investigators did not not found the in literature the study with design and calculation prediction according to the calculation of this study with the effect size of f = 0.24 for the sample calculation. Thus, was found a minimum required sample of 38 subjects (19 per group).

Results were found as mean ± standard error. Unpaired testing was used to compare baseline characteristics between groups. Comparison between groups and duration of arterial stiffness, lipid profile, glucose profile, climacteric symptoms, body composition and ABPM were made by Generalized Equation Estimates (GEE) of two factors (time, group and their interaction) with Bonferroni correction. The analyzes were performed by intention-to-treat (including those who did not complete the study: MORB n = 18; MULTI = 24) using the last-observation carried forward method. A p value <0.05 was used for statistical significance and all statistical analyzes were performed with Statistical Package for the Social Sciences (SPSS) software v26.0 (IBM, New York, USA).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (amenorrhea of at least 12 months; Estradiol <32.2 pg / mL),
* Aged between 50 and 70 years,
* Able to do aerobic exercise on track, do not have physical problems or cardiovascular complications that prevent them from exercising.
* Non-smokers ,
* Who do not use Hormone Therapy or have not finished the treatment for more than 1 year,
* As diagnostic criteria for cardiometabolic diseases: Obesity (BMI> 29.9 kg / m2; Use of antihypertensive drugs and/or hypertension (systolic blood pressure at rest > 139 mmHg and diastolic blood pressure > 89 mmHg; dyslipidemia (LDL ≥160mg / dL and / or triglycerides ≥150mg / dL and / or total cholesterol ≥190mg / dL and / or HDL ≤50mg / dL. In the case of diabetics (blood glucose > 126 mg / dL and / or HbA1c ≥ 6.5% and diagnosed with type 2 diabetes mellitus: for at least one year, being using a hypoglycemic and clinically stable for up to minimum 6 months, with glycemic control by medication or exogenous insulin and without chronic complications such as diabetic foot, nephropathy, retinopathy or neuropathies.

Exclusion Criteria:

* Present some inability to carry out the prescribed training volume or intensity,
* Not obtain medical clearance after maximum exercise test
* Start practicing another physical exercise protocol concurrently with this project.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Arterial stiffness in 12 weeks | Before and after 12 weeks of intervention
  Arterial stiffness was assessed by measuring the Pulse Wave Velocity (PWV) through the applanation tonometry method, performed on 3 measurements and the average of the three was performed to obtain the final value. It is a non-invasive, painless method with instantaneous results and considered the gold standard for determining arterial stiffness. This method is based on the principles of ocular tonometry used to measure intraocular pressure by "flattening" the surface of the eyeball.
Change in Lipid profile in 12 weeks | Before and after 12 weeks of intervention.
  The blood samples were collected after an overnight fast, five days before, and 72 h after, the last exercise training session to eliminate the acute effects of the exercise. Plasma concentrations of total cholesterol (mg/dL), triglycerides (mg/dL), high density lipoprotein (HDL) (mg/dL) and low density lipoprotein (LDL) cholesterol (mg/dL) were determined by enzymatic colorimetric methods. All analyzes were performed using an automated system using commercial kits.
Change in 24-hour ambulatory blood pressure in 12 weeks | Before and after 12 weeks of intervention.
  Blood pressure (Systolic, diastolic, mean) (mmHg) was assessed before and after 12 weeks of training through ambulatory monitoring (ABPM) using the Dyna Mapa+ device (São Paulo, Brazil). The monitor was programmed with measurements every 30 minutes for 24 hours, standardizing the start of monitoring in the morning between 7 am and 8 am. Along with the monitor, the participants filled out a daily record of activities (sleep, food and work) or events that could interfere with blood pressure or measurements, with sleep and wakefulness periods being individually determined according to the time reported in each diary. Measurements obtained 24 hours of monitoring and with at least 70% of measurements valid in this period were considered valid.
Change in glycated hemoglobin (HbA1c) | Before and after 12 weeks of intervention.
  The blood samples were collected after an overnight fast, five days before, and 72 h after, the last exercise training session to eliminate the acute effects of the exercise. The concentration (%) of glycated hemoglobin (HbA1c) was determined by the turbidimetry method. All analyzes were performed using an automated system, using commercial kits.
Change in glucose | Before and after 12 weeks of intervention.
  The blood samples were collected after an overnight fast, five days before, and 72 h after, the last exercise training session to eliminate the acute effects of the exercise. Plasma concentrations of glucose (mg/dL) were determined by enzymatic colorimetric methods. The analyze was performed using an automated system using commercial kit.

SECONDARY OUTCOMES:
Blood Pressure Variability | Before and after 12 weeks of intervention
  The systolic, diastolic and mean blood pressure values (mmHg) from the Ambulatory Blood Pressure Monitoring will be used in the assessment of Blood Pressure Variability (BPV) according to the protocols. Comparing the variables between groups: Standard deviation, Coefficient of variation, real average variability (ARV), morning surge, night descent, with individuals classified as: present, attenuated, absent or accentuated descent, when the pressure decreases between periods wakefulness and sleep is ≥ 10%, < 10%, ≤ 0%, and ≥ 20%, respectively; Percent pressure loads of systolic blood pressure values greater than 130 mmHg during the 24 hours, greater than 135 mmHg during the waking period and greater than 120 mmHg during the sleep period; and diastolic blood pressure greater than 80 mmHg during the 24 hours, greater than 85 mmHg during the waking period and greater than 70 mmHg during the sleep period.
Heart rate variability | Before and after 12 weeks of intervention
  The analysis of heart rate variability (HRV) will be analyzed in the frequency and time domain, using a specific software for such analysis. In the time domain, the following indexes will be calculated: interval between two consecutive R waves (RR), (RMSSD) square root of the mean of the sums of the squared differences of the adjacent RR intervals; (SDNN) standard deviation of all normal RR intervals in a time interval; (pNN50) Percentage of adjacent RR interval pairs that are at least 50 ms apart during recording.
  For frequency domain analysis: the series of RR intervals, to calculate the power density of the spectrum, the fast Fourier transform (FFT) will be used. The high (HF) and low (LF) frequency spectrum zones will be calculated from the integral of the spectrum power density curve in their respective zones.
Assessment of anthropometry | Before and after 12 weeks of intervention
  Anthropometric assessments were carried out in a reserved environment, in which waist, hip and abdomen circumferences (cm) were assessed using a 0.5 cm wide inelastic measuring tape device.
Assessment of climacteric symptoms - Cervantes Quality of Life Scale | Before and after 12 weeks of intervention.
  Climacteric symptoms were assessed using the Cervantes Quality of Life Scale, which has 31 questions in the domains: menopause and health, psychic domain, marital relationship and sexuality, and the score goes from 0 to 155, considering that the higher the total score, the worse the quality of life.
Change in Body composition in 12 weeks | Before and after 12 weeks of intervention.
  The assessment of body composition (kg) was performed using the Bioimpedance technique, which features a tetrapolar system with 8 electrodes and a frequency of 20-100 kilohertz.
Assessment of climacteric symptoms - Menopause Rating Scale (MRS) | Before and after 12 weeks of intervention.
  The Menopause Rating Scale (MRS) is composed of eleven questions and the symptoms are divided into somatovegetative, psychological and urogenital. Classification according to total score: asymptomatic or sparse (0-4 points), mild (5-8 points), moderate (9-15 points) or severe (more than 16 points).

CONTACTS AND LOCATIONS:
Overall Officials: Juliene Dechichi, MSc, Principal Investigator — Federal University of Uberlandia; Guilherme Puga, PhD, Study Director — Federal University of Uberlandia
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laurent S, Cockcroft J, Van Bortel L, Boutouyrie P, Giannattasio C, Hayoz D, Pannier B, Vlachopoulos C, Wilkinson I, Struijker-Boudier H; European Network for Non-invasive Investigation of Large Arteries. Expert consensus document on arterial stiffness: methodological issues and clinical applications. Eur Heart J. 2006 Nov;27(21):2588-605. doi: 10.1093/eurheartj/ehl254. Epub 2006 Sep 25. PMID 17000623
- [Background] Kario K, Matsuo T, Kobayashi H, Imiya M, Matsuo M, Shimada K. Nocturnal fall of blood pressure and silent cerebrovascular damage in elderly hypertensive patients. Advanced silent cerebrovascular damage in extreme dippers. Hypertension. 1996 Jan;27(1):130-5. doi: 10.1161/01.hyp.27.1.130. PMID 8591875
- [Background] Lima JE, Palacios S, Wender MC. Quality of life in menopausal women: a Brazilian Portuguese version of the Cervantes Scale. ScientificWorldJournal. 2012;2012:620519. doi: 10.1100/2012/620519. Epub 2012 Mar 12. PMID 22500142
- [Background] Heinemann LA, Potthoff P, Schneider HP. International versions of the Menopause Rating Scale (MRS). Health Qual Life Outcomes. 2003 Jul 30;1:28. doi: 10.1186/1477-7525-1-28. PMID 12914663
- [Background] Heinemann K, Ruebig A, Potthoff P, Schneider HP, Strelow F, Heinemann LA, Do MT. The Menopause Rating Scale (MRS) scale: a methodological review. Health Qual Life Outcomes. 2004 Sep 2;2:45. doi: 10.1186/1477-7525-2-45. PMID 15345062
- [Background] Banegas JR, Ruilope LM, de la Sierra A, Vinyoles E, Gorostidi M, de la Cruz JJ, Ruiz-Hurtado G, Segura J, Rodriguez-Artalejo F, Williams B. Relationship between Clinic and Ambulatory Blood-Pressure Measurements and Mortality. N Engl J Med. 2018 Apr 19;378(16):1509-1520. doi: 10.1056/NEJMoa1712231. PMID 29669232 (Retraction: PMID 31995856 N Engl J Med. 2020 Jan 29;382(8):786)
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Tarvainen MP, Niskanen JP, Lipponen JA, Ranta-Aho PO, Karjalainen PA. Kubios HRV--heart rate variability analysis software. Comput Methods Programs Biomed. 2014;113(1):210-20. doi: 10.1016/j.cmpb.2013.07.024. Epub 2013 Aug 6. PMID 24054542